CLINICAL TRIAL: NCT03875014
Title: Comparison of Bipolar Hemiarthroplasty and Total Hip Arthroplasty With Dual Mobility Cup in the Treatment of Old Active Patients With Displaced Neck of Femur Fracture
Brief Title: Comparison of Bipolar Hemiarthroplasty and Total Hip Arthroplasty With Dual Mobility Cup
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, shah fahad, Principal Investigator, Aga Khan University
Other Study IDs: AKUP
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Dislocations
Keywords: dual mobility cup; total hip repcament; bipolar hemiarthroplasty; dislocation
MeSH Terms: conditions — Joint Dislocations | interventions — Surgical Procedures, Operative; Mutagenesis, Insertional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: Bipolar hemiarthroplasty grop
  Interventions: Device: surgery with implant for hip fracture
- group 2: Total hip replacement dual mobility group
  Interventions: Device: surgery with implant for hip fracture

INTERVENTIONS:
Device: surgery with implant for hip fracture — hip replacement with bipolar hemiarthroplasty or total hip arthroplasty dual mobility done and patients was followed

SUMMARY:
This study is conducted with the aim to compare the functional outcome, rate of dislocation, complications and mortality after treatment of displaced neck of femur fracture with bipolar hemiarthroplasty or total hip arthroplasty with dual mobility cuff.

DETAILED DESCRIPTION:
This study is conducted with the aim to compare the functional outcome, rate of dislocation, complications and mortality after treatment of displaced neck of femur fracture with bipolar hemiarthroplasty or total hip arthroplasty with dual mobility cuff.

This study is conducted with the aim to compare the functional outcome, rate of dislocation, complications and mortality after treatment of displaced neck of femur fracture with bipolar hemiarthroplasty or total hip arthroplasty with dual mobility cuff.

A retrospective cohort study will be conducted at our tertiary care level 1 trauma center .ERC approval wwill taken from Ethical Review Committee of the hospital. Patients of age group more than 60 year who underwent hip arthroplasty (bipolar hemiarthroplasty or THA with dual mobility implant) between 2015 and 2017 for displaced neck of femur fracture with a complete follow up for one year were included.

Both groups will be assessed for postoperative complications including surgical complications (dislocation, periprosthetic fracture and surgical site infection), one year mortality and functional outcome via Harris hip score at the latest follow up.

Data will be analyzed using SPSS version 20.Chi-sqaure test was used to compare categorical variables whereas independent sample T-test was used to compare continuous variables. P-value of <0.05 was considered significant

ELIGIBILITY:
Inclusion Criteria:

* . Patients of age group more than 60 year who underwent hip arthroplasty (bipolar hemiarthroplasty or THA with dual mobility implant) between 2015 and 2017 for displaced neck of femur fracture with a complete follow up for one year

Exclusion Criteria:

* Patient who underwent hip arthroplasty for other indications, patients younger than 60 years patient with pathological fractures, patient with missing records and patients lost to follow up

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: . Patients of age group more than 60 years old with hip fracture treated via bipolar hemiarthroplasty or total hip replacement with dual mobility cup
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
mortality | one year
  death within one year of index surgery

SECONDARY OUTCOMES:
functional outcome | one year
  harris hip score used to determine functional outcome

IPD SHARING:
Plan to Share IPD: Undecided